CLINICAL TRIAL: NCT06751693
Title: Development of a Scoring and Prediction Model for Weaning Success in ARDS Patients Using Ventilation Parameters Combined with Artificial Intelligence and Deep Learning Techniques
Status: Completed | Type: Observational
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2024-12-07
Record Dates: First submitted 2024-12-11; First posted 2024-12-30 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Deep Learning; Artificial Intelegence; ARDS (Acute Respiratory Distress Syndrome)
Keywords: Deep Learning
MeSH Terms: conditions — Acute Lung Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Weaned: Those successfully weaned from mechanical ventilation
- Non-weaned: Those who not weaned from mechanical ventilation

SUMMARY:
This study aims to develop an AI-supported scoring model to optimize the weaning processes of ARDS patients from mechanical ventilation. Retrospective analysis will be conducted on the data of 25,000 patients, focusing on ventilator parameters and hemodynamic variables. The model will be designed to contribute to clinical decision support systems.

DETAILED DESCRIPTION:
The aim of this study is to develop an artificial intelligence and deep learning-supported scoring system using ventilator parameters obtained during the mechanical ventilation process in patients diagnosed with ARDS. This system seeks to predict and optimize the weaning process, facilitating successful liberation from mechanical ventilation.

In this context, our study will analyze data from 25,000 patients obtained from the Metavision system. From this data pool, ARDS patients will be filtered and divided into two groups: those successfully weaned from mechanical ventilation (weaned) and those who were not (non-weaned). The ventilator parameters of both groups, including oxygenation indices, driving pressure, and total mechanical power, will be examined in detail.

The collected data will be analyzed using artificial intelligence and deep learning algorithms to develop a scoring system capable of predicting patients' weaning processes. This system is designed to guide clinicians in patient management and enhance the success of weaning procedures.

The results of this study aim to contribute to more efficient and safer management of the weaning process for ARDS patients. Furthermore, the implementation of AI-supported scoring systems in intensive care units is expected to promote widespread adoption and improve the quality of patient care.

ELIGIBILITY:
Inclusion Criteria:

* ARDS diagnosis
* Aged 18 years and older
* Intubated and followed by Mechanical ventilation
* Admission on Intensive care unit
* Complete data on clinical support and desicion system

Exclusion Criteria:

* Missing data
* Under 18 years of age
* Followed by non-ARDS conditions
* Terminal status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intubated patients which diagnosed with ARDS and followed up in the ICU for more than 48 hours.
Sampling Method: Non-Probability Sample
Enrollment: 25000 (Actual)
Dates: Start 2024-12-10 (Actual); Primary Completion 2024-12-24 (Actual); Study Completion 2024-12-24 (Actual)

PRIMARY OUTCOMES:
Successful Weaning | 48 hours
  The primary outcome of this study will be the successful weaning from mechanical ventilation.

SECONDARY OUTCOMES:
Mechanical Ventilatory Parameters | 48 hours
  Determining the impact of mechanical power on patient outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Zafer Cukurova, M.D, Study Chair — Bakırkoy Dr. Sadi Konuk Training and Research Hospital
Locations (1):
- Bakirkoy Dr Sadi Konuk Research and Training Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No